CLINICAL TRIAL: NCT03853590
Title: Mechanisms Underlying the Improvement of Insulin Resistance in Response to Bariatric Surgery
Brief Title: Improvement of Insulin Resistance After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beth Israel Deaconess Medical Center (Other)
Responsible Party: Principal Investigator, Christos Mantzoros, Principal Investigator, Beth Israel Deaconess Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 2009P-000216
Record Dates: First submitted 2019-02-22; First posted 2019-02-25 (Actual); Last update posted 2019-02-25 (Actual); Status verified 2019-02

CONDITIONS: Obesity; Bariatric Surgery Candidate; Insulin Tolerance
MeSH Terms: conditions — Obesity | interventions — Gastric Bypass

STUDY DESIGN:
Intervention Model Description: Eligible patients were consecutively recruited and treatment allocation was decided after clinical evaluation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Laparoscopic Adjustable Gastric Band (Active Comparator): Subjects who elected to undergo Laparoscopic Adjustable Gastric Band intervention were examined prior to surgery and at 2, 3, 6 months after operation.
  Interventions: Procedure: Laparoscopic adjustable gastric banding
- Roux-en-Y gastric bypass surgery (Experimental): Subjects who elected to undergo Roux-en-Y gastric bypass surgery were examined prior to surgery and at 2, 3, 6 months after operation.
  Interventions: Procedure: Roux-en-Y gastric bypass

INTERVENTIONS:
Procedure: Roux-en-Y gastric bypass — Creation of a small pouch from the stomach and connection of the newly created pouch directly to the small intestine so that swallowed food bypasses most of the stomach and the first section of the small intestine.
  Arms: Roux-en-Y gastric bypass surgery
Procedure: Laparoscopic adjustable gastric banding — Placement of a soft silicone ring with an expandable balloon in the center, around the top part of the stomach to create a two-compartment stomach, with a much smaller top part above the band. The subject will eat enough food only to fill the top part of the stomach decreasing caloric consumption.
  Arms: Laparoscopic Adjustable Gastric Band

SUMMARY:
Non-randomized open label study to investigate factors mediating changes in insulin sensitivity, glucose tolerance and other metabolic outcomes after bariatric surgery.

DETAILED DESCRIPTION:
Bariatric and weight loss surgery is an effective treatment for severe obesity. Bariatric surgery also decreases insulin resistance and improves diabetes. Our study enrolled individuals approved for bariatric surgery to collect data on modifiable predictors and laboratory outcomes. These data would allow us to systematically assess clinical outcomes over one year post bariatric surgery and elucidate how insulin resistance is decreased and diabetes is improved.

The type of surgery was selected by the subjects between Roux-en-Y gastric bypass or a laparoscopic adjustable gastric banding. Participation in the study involved having a small sample of tissue obtained from the abdomen and subjects were also given the option to have a biopsy performed in the thigh area during their elective surgical procedure (optional adipose and muscle tissue biopsies).

Subjects were examined prior to surgery and at 2, 3, 6 months after intervention. Anthropometric and body composition measurements were performed using the Bioelectrical Impendence Analysis (BIA) before surgery and 6 months post operatively. Morning blood was collected after overnight fasting during each visit. Some of the non-diabetic subjects completed a mixed nutrient stimulation study during the baseline and 6-month visit. Blood samples were collected immediately prior to drinking the liquid drink, and every 30 minutes after the meal ingestion for 2 hours.

ELIGIBILITY:
Inclusion Criteria:

1. males and females
2. 18-65 years old
3. approved for bariatric surgery as per BIDMC Bariatric Clinic guidelines
4. English-speaking
5. willing and able to take part in a multi year study involving telephone interviews and enrolled prior to bariatric surgery

Exclusion Criteria:

1. Any condition that would exclude a patient from bariatric surgery as listed below:

   1. patients with untreated major depression or psychosis
   2. binge eating disorders
   3. current drug and alcohol abuse
   4. severe cardiac disease with prohibitive anesthetic risks
   5. severe coagulopathy
   6. inability to comply with nutritional requirements including life-long vitamin replacement.
   7. pregnancy
2. Any additional condition not in accordance with standard of care as per Bariatric Clinic at BIDMC.
3. Any condition which in the opinion of the investigators rendered the candidate unsuitable for participation in this study.

Exclusion Criteria for Optional Biopsy:

1. history of any illness, other than obesity, that may affect insulin sensitivity (diabetes anemia, infectious diseases, renal or hepatic failure, uncontrolled hypertension, cancer or lymphoma)
2. subjects who required special diet prior to surgery
3. chronic inflammatory conditions such as inflammatory bowel disease and rheumatoid arthritis
4. states of cortisol or growth hormone excess
5. any medications that are known to influence glucose metabolism such as glucocorticoids
6. a known history of anaphylaxis or anaphylactoid-like reactions or who have a known hypersensitivity to anesthetic agents such as Lidocaine or Novocaine
7. a known history of bleeding dyscrasia or poor wound healing
8. any medical condition precluding supine position

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2010-02-25 (Actual); Primary Completion 2013-04-01 (Actual); Study Completion 2015-05-01 (Actual)

PRIMARY OUTCOMES:
fasting insulin | Change from Baseline insulin at 6 months post-surgery
  circulating levels of fasting insulin measured in pmol/L
fasting glucose | Change from Baseline insulin at 6 months post-surgery
  circulating levels of fasting glucose measured in mg/dl
Boost Challenge Test | Change from Baseline insulin at 6 months post-surgery
  serum insulin and glucose levels after a mixed meal challenge (Boost Protein shake)

CONTACTS AND LOCATIONS:
Overall Officials: Christos Mantzoros, MD, PhD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No